CLINICAL TRIAL: NCT05814458
Title: The Efficiency of Transcranial Direct Current Stimulation in the Treatment of Anorexia Nervosa - a Randomised, Double-blind Clinical Trial
Brief Title: The Efficiency of Transcranial Direct Current Stimulation in the Treatment of Anorexia Nervosa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/24/01/2022
Record Dates: First submitted 2023-01-31; First posted 2023-04-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Brain stimulation; Eating disorders; Left dorsolateral prefrontal cortex; Transcranial direct current stimulation
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Active Comparator): The tDCS group will receive the active brain stimulation.
  Interventions: Device: tDCS
- Placebo group (Sham Comparator): The placebo group will receive the sham brain stimulation.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: tDCS — Patients will be receiving twice a day tDCS (applied current at 2mA) stimulation, for 3 weeks on working days (30 sessions in total) and each stimulation will last 25 minutes. The anode will be located on the left, while the cathode- on the right dorsolateral prefrontal area of scalp. The commercially available Soterix 1x1 tDCS mini-CT LTE device (model 1601-LTE) will be used for stimulation.
  Arms: tDCS group
Device: Placebo — Patients will be receiving twice a day sham stimulation, for 3 weeks on working days (30 sessions in total) and each stimulation will last 25 minutes. The anode will be located on the left, while the cathode- on the right dorsolateral prefrontal area of scalp. The commercially available Soterix 1x1 tDCS mini-CT LTE device (model 1601-LTE) will be used for stimulation.
  Arms: Placebo group

SUMMARY:
The main goal of the study (a 3-week, randomized, double-blind, and placebo-controlled study) is to determine the effect of Transcranial Direct Current Stimulation (tDCS) on the mental state and advances in nutritional rehabilitation in patients with AN. The primary hypothesis assumes that tDCS will reduce the symptoms of depression, improve cognition functions and it will have a positive effect on the reduction of restriction related to body weight and diet.

DETAILED DESCRIPTION:
The aim of the study is to assess the effect of tDCS stimulation on psychological and biological factors in patient suffering for AN with particular attention to the safety of such additional therapy. Transcranial direct current stimulation (tDCS) is a non-invasive and currently considered safe method of neurostimulation. It is based on the use of direct current of very low intensity, up to 2000uA-2mA, and supplying it to the brain through electrodes placed on the scalp. In this way, the polarity of the cell membranes of neurons is induced, and this influences changes in the cortical excitation of the brain.

Results confirming the efficacy of such a therapeutic approach would provide support for the introduction of brain stimulations as a valuable part of treatment in psychiatric wards but also as a part of home-based treatment.

The protocol was developed by a multidisciplinary researcher team of a psychiatrist, psychologist, psychotherapist and nutritionists. Thanks to this, it is possible to evaluate the progress taking place in various fields.

To the best of our knowledge, this will be the first intervention study assessing the efficacy of tDCS in AN taking into account not only psychological tests, but also biochemical markers (including levels of neurotrophins) or the electrical activity of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Signed written Informed Consent Form,
* Patients aged 10-30 years old,
* Meet the DSM-5 criteria for AN,
* Body mass index (BMI) ≤ 17,5 kg/m2,
* A willingness and motivation to follow the study protocol.

Exclusion Criteria:

* Not giving Informed, Written Consent
* Diagnosis of neurological diseases, as epilepsy;
* Contraindications to tDCS, ie. pacemakers, metal parts around the head;
* Psychiatric comorbidities (except specific personality disorder) including mental retardation, organic brain dysfunction, or addiction (except nicotine and caffeine);
* Pregnancy or pregnancy planning;
* Changes in psychopharmacotherapy during hospitalization

Ages: 10 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in severity of eating disorder symptoms 1 | The test will be performed four times: Before stimulation, baseline (V1), immediately after stimulation (V2) two weeks after the intervention (V3), and two months after the intervention (V4)
  The severity of symptoms will be assessed with Eating Attitudes Test (EAT-26)
Change in severity of eating disorder symptoms 2 | The test will be performed three times: Before stimulation, baseline (V1), immediately after stimulation (V2) and two weeks after the intervention (V3)
  The severity of symptoms will be assessed with Eating Disorder Examination Questionnaire (EDE-Q 6.0).
Change in eating habits and opinions about food and nutrition | The test will be performed two times: Before stimulation, baseline (V1) and two weeks after intervention (V3)
  To evaluate changes in eating habits and opinions about food and nutrition the Questionnaire of Eating Behaviours (QEB) will be used. It is a qualitative questionnaire designed to study eating habits and opinions about food and nutrition. The first part of the questionnaire covers the frequency of consumption of selected products, the frequency of eating meals and their typical composition. In the second part of the questionnaire, there are 26 statements about food and nutrition, which enable the assessment of the level of nutritional knowledge of the respondents.
Change in food intake variety | The test will be performed three times: Before stimulation, baseline (V1), immediately after stimulation (V2) and two weeks after the intervention (V3)
  Food Intake Variety will be assessed with The Variety Food Consumption Questionnaire. It is a qualitative food consumption frequency questionnaire. It is a simple tool to collect information on the consumption of (yes / no) 63 assortment groups of products.
Change in assessment of stress levels | The test will be performed four times: Before stimulation, baseline (V1), immediately after stimulation (V2) two weeks after the intervention (V3), and two months after the intervention (V4)
  The severity of stress will be assessed with Perceived Stress Scale (PSS-10). This test consists 10 questions and is used to measure stress based on subjective feelings related to problems and personal events, behavior, coping with stress.
Change in severity of depressive symptoms 1 | The tests will be performed twice: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  Severity of depressive symptoms will be assessed with Beck's Depression Inventory (BDI)
Change in severity of depressive symptoms 2 | The tests will be performed three times: Before stimulation, baseline (V1), immediately after stimulation (V2), and two months after the intervention (V4)
  Severity of depressive symptoms will be assessed with Questionnaire for the Diagnosis of Depression in Children and Adolescents (CDI2).
Change in meta-cognition | The test will be performed three times: Before stimulation, baseline (V1), immediately after stimulation (V2), and two months after the intervention (V4)
  To assess metacognitive abilities Meta-Cognition Questionnaire (MCQ-A) will be used. Reliable and valid instrument for measuring meta-cognitive beliefs in adolescents (12-18 lat). The MCQ-A assesses the severity of dysfunctional meta-cognitive beliefs in adolescents (12-18) that affect their daily functioning. The first and second subscales measures "positive and negative beliefs about worry," Subscale 3 measures "cognitive confidence," Subscale 4 measures "beliefs about superstition, punishment and responsibility". Finally, subscale 5 measures "cognitive self-consciousness,".
Change in attention and perceptiveness | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To assess levels of attention Color connection test (CTT-1, CTT-2) and Test of attention and perceptiveness will be used.
Change in intensity of intrusive thoughts | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To assess intensity of intrusive thoughts CY-BOCS scale will be used
Change in intensity of rumination | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To assess intensity of rumination the Ruminance-Reflectivity Questionnaire will be used
Change in visual memory | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To assess visual memory test BENTON will be used. This test is used to test memory, visual perception and graphomotor skills. The examined person draws the presented patterns (10 pieces) from memory or redraws them, depending on the version and methods of the research carried out by the researcher.
Change in body image self-esteem | The test will be performed three times: Before stimulation, baseline (V1), immediately after stimulation (V2) and two weeks after the intervention (V3)
  To assess body image self-esteem Appearance Self-Rating Sheet (ASRS) will be used. Assessment of 25 dimensions related to your body - (different parts of your body). The patient receives a visualization of the body figure on the drawing and evaluates its individual elements. The test allows you to assess the importance of appearance for patients, the assessment of satisfaction with one's appearance and the satisfaction index. The SES self-assessment questionnaire will also be used
Change in cognitive abilities 1 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To assess cognitive abilities Matching Familiar Figures Test (MFF)
Change in cognitive abilities 2 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To assess cognitive abilities Verbal Fluency Test will be used.
Change in self-esteem | The test will be performed three times: Before stimulation, baseline (V1), immediately after stimulation (V2) and two weeks after the intervention (V3)
  The Rosenberg Self-Esteem Scale (SES) will be used. SES is a tool for assessing the level of general self-esteem - a relatively stable disposition understood as a conscious attitude (positive or negative) towards the Self
Change in emotion regulation | The test will be performed three times: at baseline (V1), immediately after stimulation (V2), and 2 months after stimulation (V4).
  A shortened 16-item version of a questionnaire designed for the rapid assessment of difficulties in emotion regulation Difficulties in Emotion Regulation Scale DERS-16 wil be performed. The scale measures five domains, such as lack of emotional acceptance, impulsivity, and difficulties with goal-directed behavior, using a 5-point scale.
Change in autistic traits | The test will be administered three times: at baseline (V1), immediately after stimulation (V2), and 2 months after stimulation (V4).
  The Autism Spectrum Quotient (AQ) is a self-administered questionnaire used to measure the degree to which a person shows autistic traits.
Change in mental states | The test will be administered three times: at baseline (V1), immediately after stimulation (V2), and 2 months after stimulation (V4).
  The questionnaire Mentalization Scale (MentS) is used for a rapid assessment of the capacity to reflect on mental states (emotions, intentions, and beliefs).
Change in body-related conversations | The test will be peformed three times: at baseline (V1), immediately after stimulation (V2), and 2 months after stimulation (V4).
  Family Talk Questionnaire Fat Talk refers to negative, body-related conversations between girls or young women.
Change in cognitive functions | The test will be performed twice: at baseline (V1), immediately after stimulation (V2)
  A neuropsychological diagnostic tool Rey-Osterrieth Complex Figure used to assess visuospatial abilities, visual memory, and executive functions (planning and organization).
Change in anxiety level | The test will be performed three times: at baseline (V1), immediately after stimulation (V2), and 2 months after stimulation (V4).
  The STAI (State-Trait Anxiety Inventory) is a psychological tool used to measure anxiety as both a state (a temporary feeling of tension) and a trait (a stable personality disposition). It consists of two subscales (X-1 and X-2, or Y-1 and Y-2), each containing 20 questions, with scores ranging from 20 to 80 points.

SECONDARY OUTCOMES:
Change in electrolyte levels | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate electrolyte levels (mmol/l) in blood serum following tests will be performed:
  sodium, phosphorus, magnesium, calcium, potasium
Change in morphotic elements 1 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  RBC - Red Blood Cell (M/µl)
Change in morphotic elements 2 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  Hemoglobin (mmol/l) Mean Corpuscular Hemoglobin Concentration (mmol/l)
Change in morphotic elements 3 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  Hematocrit
Change in morphotic elements 4 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  Mean Corpuscular Volume (fl)
Change in morphotic elements 5 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  Mean Corpuscular Hemoglobin (pg)
Change in morphotic elements 6 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  Ferritin ( ng/ml)
Change in morphotic elements 7 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  White Blood Cell (K/µl) Lymphocytes (K/µl)
Change in morphotic elements 8 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate morphotic elements complete morphology with smear will be performed:
  Monocytes (G/l)
Metabolic changes 1 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate metabolic changes in blood serum Thyroid parameters will be examined: FT3 (pmol/l), FT4 (pmol/l)
Metabolic changes 2 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate metabolic changes in blood serum the pituitary gland parameter will be examined: TSH (µIU/ml)
Neurophysiologic changes 1 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate neurophysiologic changes EEG (theta and alpha wave power) test will be performed
Change in neurotrophin levels | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate neurotrophin levels in blood serum tests will be performed: BDNF (pg/ml), Neurotrphin 3 and 4 (pg/ml), NGF (pg/ml)
Change in food intake regulators: | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate food intake regulators in blood serum tests will be performed: leptin (pg/ml), visfatin (pg/ml)
Body composition changes 1 | The test will be performed four times: Before stimulation, baseline (V1), immediately after stimulation (V2), two weeks after the intervention (V3), and two months after the intervention (V4)
  To evaluate body composition changes BIA body composition analysis will be performed: Body weight (kg)
Body composition changes 2 | The test will be performed four times: Before stimulation, baseline (V1), immediately after stimulation (V2), two weeks after the intervention (V3), and two months after the intervention (V4)
  To evaluate body composition changes BIA body composition analysis will be performed: Intracellular and extracellular water (l/%)
Body composition changes 3 | The test will be performed four times: Before stimulation, baseline (V1), immediately after stimulation (V2), two weeks after the intervention (V3), and two months after the intervention (V4)
  To evaluate body composition changes BIA body composition analysis will be performed: Lean body mass (kg/%)
Body composition changes 4 | The test will be performed four times: Before stimulation, baseline (V1), immediately after stimulation (V2), two weeks after the intervention (V3), and two months after the intervention (V4)
  To evaluate body composition changes BIA body composition analysis will be performed: Fat mass (kg/%)
Changes in HPA axis biomarker | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate HPA axis cortisol (nmol/l) in blood serum will be tested
Metabolic changes 3 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate metabolic changes in blood serum Total Protein parameter will be examined.
Metabolic changes 4 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate metabolic changes in blood serum the glucosis level will be performed.
Cardiac Parameter Changes | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate changes in cardiac parameters in blood serum, NT-proBNP will be measured (pg/mL).
Metabolic changes 5 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate metabolic changes in blood serum, a lipid profile parameter will be measured: total cholesterol (mg/dL)
Metabolic changes 6 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2).
  To evaluate metabolic changes in blood serum, a lipid profile parameter will be measured: LDL cholesterol (mg/dL).
Metabolic changes 7 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2).
  To evaluate metabolic changes in blood serum, a lipid profile parameter will be measured: triglycerides (mg/dL).
Metabolic changes 8 | The test will be performed two times: Before stimulation, baseline (V1) and immediately after stimulation (V2)
  To evaluate metabolic changes in blood serum, a lipid profile parameter will be measured: non-HDL cholesterol (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Karakuła-Juchnowicz, Prof., Study Director — 1st Department of Psychiatry, Psychotherapy and Early Intervention, Medical University of Lublin
Locations (1):
- Ist Department of Psychiatry, Psychotherapy and Early Intervention, Lublin, Lublin Voivodeship, Poland

REFERENCES:
- [Derived] Rzad Z, Rog J, Kajka N, Szewczyk P, Krukow P, Karakula-Juchnowicz H. The efficacy of transcranial direct current stimulation in the treatment of anorexia nervosa: a randomized double-blind clinical trial. Front Psychiatry. 2024 May 2;15:1284675. doi: 10.3389/fpsyt.2024.1284675. eCollection 2024. PMID 38757134